CLINICAL TRIAL: NCT01485653
Title: Effective Low Dosage of Mepivacaine in Ultrasound Guided Axillary Block in Patients Undergoing Distal Upper Extremity Surgery
Brief Title: Dosage of Mepivacaine in Ultrasound Axillary Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Samuel Perov, Dr Samuel Perov, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: WSU irb# 0902006824; need to get (Other: WSU IRB)
Record Dates: First submitted 2011-11-23; First posted 2011-12-05 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Nerve Block; Neuromuscular Blockade; Anesthesia
Keywords: Brachial Plexus; Mepivacaine; Ultrasound; Axillary; Block
MeSH Terms: conditions — Bites and Stings | interventions — Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepivacaine, Ultrasound Axillary Block (Experimental): Group 1) 20mL 1.5% mepivacaine Group 2) 30mL 1.5% mepivacaine
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Drug: Mepivacaine — Group 1) 20mL 1.5% mepivacaine, one dose Group 2) 30mL 1.5% mepivacaine, one dose

SUMMARY:
The use of ultrasonography as an adjunct to regional anesthesia has significantly increased in recent years. Brachial plexus blockade by an axillary approach is amenable to the use of ultrasound guidance. Real time sonography of nerve structures ensures an optimal distribution of the block solution. When compared to other methods of nerve localization, sonography decreases: failure rate procedure time and the onset time for blockade. Furthermore, the use of ultrasound for peripheral nerve blockade demonstrates decreased procedure related complications such as nerve injury and unintentional vascular puncture.

Traditional axillary block techniques relying on surface anatomical landmarks require large volumes of local anesthetic, generally 40mL and greater. Utilizing the increased accuracy offered by ultrasound, some studies have shown that low volumes of local anesthetic can yield successful axillary plexus blockade. Therefore, the tradition of using large volumes of local anesthetic for axillary blocks, even without ultrasound, may not be warranted.

Although recent investigations support using a low volume of local anesthetic for brachial plexus blockade, there is a lack of outcome data from blinded randomised trials. The primary objective of this study was to evaluate 2 different volumes of local anesthetic for axillary blockade: 1) 20mL or 2) 30 mL. For the 2 different volumes used in this study, a 1.5% solution of mepivacaine was chosen due to its widespread clinical use in axillary blocks, which is secondary to: rapid onset of action, intermediate duration of effect, and relative low cost. The primary outcome was block success rate for outpatients undergoing distal upper limb surgery. Secondary objectives included comparing the 2 volumes with respect to: time required to perform the block, and onset of sensory and motor blockade.

DETAILED DESCRIPTION:
Introduction

The use of ultrasonography as an adjunct to regional anesthesia has significantly increased in recent years. Brachial plexus blockade by an axillary approach is amenable to the use of ultrasound guidance. Real time sonography of nerve structures ensures an optimal distribution of the block solution. When compared to other methods of nerve localization, sonography decreases: failure rate procedure time and the onset time for blockade. Furthermore, the use of ultrasound for peripheral nerve blockade demonstrates decreased procedure related complications such as nerve injury and unintentional vascular puncture.

Traditional axillary block techniques relying on surface anatomical landmarks require large volumes of local anesthetic, generally 40mL and greater. Utilizing the increased accuracy offered by ultrasound, some studies have shown that low volumes of local anesthetic can yield successful axillary plexus blockade. Therefore, the tradition of using large volumes of local anesthetic for axillary blocks, even without ultrasound, may not be warranted.

Although recent investigations support using a low volume of local anesthetic for brachial plexus blockade, there is a lack of outcome data from blinded randomised trials. The primary objective of this study was to evaluate 2 different volumes of local anesthetic for axillary blockade: 1) 20mL or 2) 30 mL. For the 2 different volumes used in this study, a 1.5% solution of mepivacaine was chosen due to its widespread clinical use in axillary blocks, which is secondary to: rapid onset of action, intermediate duration of effect, and relative low cost. The primary outcome was block success rate for outpatients undergoing distal upper limb surgery. Secondary objectives included comparing the 2 volumes with respect to: time required to perform the block, and onset of sensory and motor blockade.

Methods

This pilot study was a prospective, double blinded, randomized trial of 64 patients recruited from the Detroit Receiving Hospital, Detroit, MI. All patients were scheduled to undergo upper limb surgery in an outpatient setting. Upon obtaining written informed consent, patients were randomly assigned to receive either 20mL (n=31) or 30mL (n=33) of a 1.5% mepivacaine solution for axillary plexus blockade. All anesthetic blocks were placed using standard medical protocol. Nerve localization was performed using a GE LOGIQe ultrasound machine (GE Medical systems, Milwaukee, Wis, USA), with a 12L-RS transducer (42mm x 7mm footprint, 5-13 MHz). Following identification of the axillary neurovascular bundle, a 22G x 50 mm poly medic UPC electric stimulation needle was inserted and advanced along the longitudinal axis of the ultrasound transducer so that the entire shaft and tip could be visualized. A peri-arterial injection of 1.5% mepivacaine in the vicinity of the individual nerve sheaths was performed after negative aspiration. The end point being the circumferential "donut sign" spread around the artery. Additionally, the musculocutaneous nerve was identified and 1.5% mepivacaine was injected around the nerve. Depending on the patient group allocation either 20mL or 30 mL total of 1.5% mepivacaine was infiltrated. For the group receiving 20mL, 15 of the total 20 mL was spread around the axillary artery and 5mL spread around the musculocutaneous nerve. For the group receiving 30mL, 20 of the total 30 mL was spread around the axillary artery and 10mL was spread around the musculocutaneous nerve. By instituting this injection technique, results could be extrapolated to non ultrasound guided axillary blocks.

Inclusion Criteria All subjects recruited into the study were patients undergoing forearm, wrist, or hand surgery, in an outpatient setting. Other attributes included: ASA I-III, BMI < 35, and age between 18-89 years. All subjects had no history of: CVA, diabetes, anxiety disorder, obstructive sleep apnea, previous surgery or scarring in the axillary to elbow area, neurological impairment of either upper extremity, allergies to local anesthesia, coagulopathy, infection at site of block, chronic opioid therapy for chronic pain, casts or dressing on the limb that would impair assessment of blocks. Pre-block sedation using < 0.8mg/kg midazolam and no administration of preoperative opioids. Block procedure time < 10min. Subjects consented to light intraoperative sedation.

Data collection Preoperatively: Demographics, ASA (marker for surgical risk), height, weight, surgical procedure, location of procedure (hand, wrist, forearm), sedation used in preoperative holding area, the amount of versed used, block start and end time (duration of time taken between needle insertion and extraction), onset of sensory blockade, onset of motor blockade.

Intraoperatively: Conversion to general anesthesia, use of local anesthesia intraoperatively, total amount of propofol administered, surgical incision time, surgery end time.

Postoperative: Complications related to axillary block. Discharge criteria met.

Onset of Sensory blockade: Examined every 5 minutes following needle extraction using a blunt needle at 4 specific anatomic locations corresponding to radial, ulnar, median, and musculocutaneous distributions and compared with contralateral side using same stimulus. Normal pinprick sharp, 3; pinprick felt but not as sharp, 2; pressure felt but no pinprick felt, 1; no sensation at all, 0.

Onset of Motor Blockade: Examined every 5 minutes following needle extraction. Wrist flexion: median nerve; wrist extension: radial nerve; abduction of 5th finger or straight finger adduction: ulnar nerve; elbow flexion (with forearm supinated): musculocutaneous nerve. Normal strength, 3; decreased strength but moves against gravity or some resistance, 2; no movement against gravity or twitch, 1; no movement at all, 0.

Definitions of successful block Functional successful block: Sensory score of 0-1 in all 4 territories and motor score of 0-1 in 3 of 4 territories within 30 minutes of needle extraction.

Surgical successful block: no required intraoperative supplemental local anesthetic, light sedation <25mcg/kg/min propofol and absence of general endotracheal anesthesia.

Statistics

An unpaired students-t-test procedure (two-sample assuming equal variances, two-tail significance p<0.05, 95% confidence interval) was performed to examine mean differences between the 2 study groups on all continuously scaled variables. A repeated measures ANOVA was used to measure differences between both groups over time for motor and sensory nerve block scores at the 6 measured time points (5 min, 10 min, 15 min, 20min, 25 min and 30 min). Assumptions of normality and/or homogeneity of variance were checked and verified. Comparisons between study groups on proportional differences were examined using a non-parametric Fisher's Exact Chi-square test, when applied to 2x2 and 2x3 tables. Statistical significance was set at a p-value ≤0.05. All continuous data is expressed as mean with 95% upper and lower confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic forearm, wrist and hand surgery
* ASA I-III
* block procedure time less than 6 minutes
* pre-block sedation using less than 2 mcg fentanyl and less than .04 mg midazolam,
* patient consent to light pre-op sedation

Exclusion Criteria:

* Elbow/arm surgery longer than 2 hours
* ASA IV
* BMI greater than 35
* Pregnant patients
* history of CVA or scarring in the axillary to elbow area
* history of neurological impairment of either upper extremity
* Any allergies to local anesthetics coagulopathy,
* infection at the site of block
* patients requiring opioid therapy for chronic pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Successful Block | 30 minutes
  Definitions of successful block Functional successful block: Sensory score of 0-1 in all 4 territories and motor score of 0-1 in 3 of 4 territories within 30 minutes of needle extraction.
  Surgical successful block: no required intraoperative supplemental local anesthetic, light sedation <25mcg/kg/min propofol and absence of general endotracheal anesthesia.

SECONDARY OUTCOMES:
Time required until onset of sensory blockade. | 30 minutes
  Onset of Sensory blockade: Examined every 5 minutes following needle extraction using a blunt needle at 4 specific anatomic locations corresponding to radial, ulnar, median, and musculocutaneous distributions and compared with contralateral side using same stimulus.
  Onset of Motor Blockade: Examined every 5 minutes following needle extraction. Wrist flexion: median nerve; wrist extension: radial nerve; abduction of 5th finger or straight finger adduction: ulnar nerve; elbow flexion (with forearm supinated): musculocutaneous nerve.
Time taken until Onset of Motor Blockade | 30 minutes
  Onset of Motor Blockade: Examined every 5 minutes following needle extraction. Wrist flexion: median nerve; wrist extension: radial nerve; abduction of 5th finger or straight finger adduction: ulnar nerve; elbow flexion (with forearm supinated): musculocutaneous nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Perov, M.D., Principal Investigator — Wayne State University, Department of Anesthesiology